CLINICAL TRIAL: NCT06659822
Title: Responding to Elder Abuse in GERiAtric Care (REAGERA) - Dementia Validation of Screening Instruments to Detect Abuse of Persons With Dementia
Brief Title: Responding to Elder Abuse in GERiAtric Care - Dementia
Acronym: REAGERA
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Collaborators: Linkoeping University (Other Government); Jonkoping County Hospital (Other); Jonkoping University (Other)
Responsible Party: Principal Investigator, Johanna Simmons, Principal Investigator, Region Östergötland
Other Study IDs: 2021-05822-01; 20210151 (Other Grant/Funding Number: Kamprad Family Foundation for Entrepreneurship, Research and Charity); 941250 and 981144 (Other Grant/Funding Number: Medical Research Council of Southeast Sweden)
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-01

CONDITIONS: Elder Abuse; Dementia
Keywords: Validation of screening instruments to detect elder abuse
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- People with dementia: People diagnosed with dementia
- Next of kin: Next of kin to people with dementia

SUMMARY:
Abuse of older people is common and people with dementia are especially susceptible to abuse. Older people may be subjected to physical, psychological, sexual, financial abuse or neglect by relatives as well as health and social care professionals or other people in a relationship involving an expectation of trust. Reporting experiences of abuse is associated with poor health outcomes. Still, abusive experiences are often unknown to professionals.

This study protocol describes the development and procedure to test the validity of two new screening instruments (REAGERA-S20 and REAGERA-N) to detect abuse of people with dementia. The aims of the study are:

1. To assess the validity of two new self-administered screening tools to detect abusive experiences among people with dementia: the REAGERA-S20 directed at people with dementia and the REAGERA-N directed at the next of kin.
2. To translate and validate a Swedish version of the Risk of Elder Abuse and Mistreatment Instrument (REAMI) that can be used by professional caregivers to estimate risk of maltreatment and abuse of people with dementia.
3. To explore experiences of abuse among people with dementia and their next of kin.

Method People with mild to moderate dementia (n=80) and their next of kin (n=80) are recruited at health and social care facilities providing care to people with dementia. In cases of severe dementia or when the person with dementia is excluded for other reasons, only next of kin is included.

The following steps are used in the data collection

1. Participants fill out the REAGERA-S20 or REAGERA-N individually.
2. Participants are interviewed individually by two different researchers about their abusive experiences. If a participant talks about abusive experiences, a qualitative in-depth interview about those experiences is conducted.
3. A preliminary classification of the participants as abused or not abused, based only on information provided in the individual interview is made.
4. Information provided in the two individual interviews are compared by the researchers. If needed, and with permission obtained individually from the participants, a joint concluding interview is conducted to clarify inconsistencies.
5. A final classification of participants experiences of abuse is made based on the information provided in both interviews.

The validity of the REAGERA-S20/REAGERA-N will be calculated using the following classification of participants made in the interviews as gold standard (aim 1):

For the person with dementia

* Reporting or not reporting abusive experiences during the past 12 months.
* Reporting or not reporting abusive experience earlier in life, i.e. more than 12 months ago.

For the next of kin

* Reporting or not reporting own exposure to abuse by the person with dementia during the past 12 months.
* Reporting or not reporting own perpetration of abuse towards the person with dementia during the past 12 months.
* Reporting or not reporting that the person with dementia has been exposed to abuse by another person during the past 12 months.
* Reporting or not reporting that the person with dementia has been exposed to abuse earlier in life, i.e. more than 12 months ago.

After completion of data collection, the REAMI is filled out by a health or social care professional with knowledge about the participant with dementia. Validity of the instrument will be calculated using the information provided in the interview as the gold standard (aim 2).

All interviews are recorded and transcribed verbatim. Analyses of the qualitative interviews will be made to explore experiences of abuse among participants (aim 3).

ELIGIBILITY:
Inclusion Criteria:

* Patient: Being diagnosed with dementia of mild to moderate degree (assessed by the Global Deterioration Scale (GDS) level 4 or 5)
* Next of kin: Being the next of kin to a person with dementia, GDS = 4-7

Exclusion Criteria:

* Both patient and next of kin: Severe psychiatric disorder, not being able to answer the questionnaires or participate in an interview, e.g. due to insufficient proficiency in Swedish, aphasia, hearing loss or similar.
* People with dementia: experiencing symptoms that may be exacerbated by study participation or make results less reliable (e.g. paranoia).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: - Patient and next of kin that come in contact with memory clinics or in muncipality care provided to people with dementia in the participating study locations.
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2025-04-09 (Actual); Study Completion 2025-04-09 (Actual)

PRIMARY OUTCOMES:
Validity of REAGERA-S20 and REAGERA-N | Participant fill out questionnaire (REAGERA-S20/REAGERA-N) at enrollment Semi-structured interview used as gold standard is conducted immediately afterwards.
  Sensitivity, specificity, positive and negative likelihood ratio as well as positive and negative predictive value of REAGERA-S20 and REAGERA-N will be calculated. The final classification made after interviewing both the person with dementia and the next of kin will be used as the gold standard.
Predictive value of the introductory screening questions in part one | Participant fill out questionnaire (REAGERA-S20/REAGERA-N) at enrollment. Semi-structured interview used as gold standard is conducted immediately afterwards.
  Test the predictive value of the introductory screening questions in part one of each instrument to identify abusive experiences as identified in part two of the instruments as well as in the final classification made after both individual and joint interview.
Validity of the REAMI | Semi-structured interview used as gold standard is conducted at enrollment. Health and social care professionals fill out the REAMI at some point between patient enrollment and end of study, but usually within a few weeks of enrollment.
  Health and social care professionals fill out the REAMI questionnaire assessing risk of abuse. Sensitivity, specificity, positive and negative likelihood ratio as well as positive and negative predictive value will be calculated for REAMI concerning its ability to detect abusive experiences. The interview conducted with participants will be used as the gold standard for calculations.

SECONDARY OUTCOMES:
Validity of REAGERA-S20 and REAGERA-N using individual interview as gold standard | Participant fill out questionnaire (REAGERA-S20/REAGERA-N) at enrollment. Semi-structured interview used as gold standard is conducted immediately afterwards.
  Sensitivity, specificity, positive and negative likelihood ratio as well as positive and negative predictive value for REAGERA-S20/REAGERA-N using only information given in the individual interview with the person with dementia or the next of kind respectively as the gold standard.
Expected associations with established outcomes (FAQ) | Participant fill out questionnaire (REAGERA-S20/REAGERA-N) as well as the FAQ at enrollment.
  Associations between reporting abuse in REAGERA-S20/REAGERA-N and high score on the Functional Activities Questionnaire (FAQ) will be calculated. The FAQ consists of ten items and each item can be scored from 0 (no dependence) to 3 (totally dependent). A sum score (0-30) will be calculated and a higher score indicates a greater dependence on others for activities in daily living.
Expected associations with established outcomes (ZBI) | Participant fill out questionnaire (REAGERA-S20/REAGERA-N) as well as the ZBI at enrollment
  Associations between reporting abuse in REAGERA-S20/REAGERA-N and high score on the Zarit Burden Interview (ZBI). The 12 items ZBI is used and each item is answered on a scale from 0 (never) to 4 (almost always). A sum score will be created for all items (range 0-48) and a higher sum score indicate a greater care giver burden.

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - Region Jönköpings Län, Jönköping
  - Region Östergötland, Linköping

IPD SHARING:
Plan to Share IPD: Yes
Anonymous quantitative data will be made available from the researcher upon reasonable request.

REFERENCES:
- [Derived] Simmons J, Floberg E, Casselgren C, Westerlind B, Sandberg J, Swahnberg K, Nagga K, Ludvigsson M, Johansson L. REAGERA-dementia: study protocol for the validation of screening instruments to detect abuse of people with dementia. BMC Geriatr. 2025 Aug 25;25(1):660. doi: 10.1186/s12877-025-06291-z. PMID 40855257
- See also: Webpage of research program — https://liu.se/en/research/reagera